CLINICAL TRIAL: NCT02752230
Title: Comparison of Exparel (Bupivacaine Liposome) to Marcaine (Bupivacaine) in Post-Surgical Analgesia for Laparoscopic Trocar Site Incisions in Bariatric Surgery
Brief Title: Comparison of Exparel to Marcaine in Post-Surgical Analgesia in Bariatrics
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Attending physician left network
Sponsor: Kettering Health Network (Other)
Responsible Party: Principal Investigator, Lauren Smith, Resident, Kettering Health Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 717168-2
Record Dates: First submitted 2016-03-31; First posted 2016-04-26 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Post Operative Pain
Keywords: Post operative pain; Bariatric Surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exparel (Bupivicaine Liposome) (Active Comparator): Patient will have Exparel (Bupivicaine Liposome) injected at Laparoscopic Port sites during the Laparoscopic Roux en Y or Laparoscopic Sleeve Gastrectomy.
  Interventions: Procedure: Laparoscopic Roux en Y gastric bypass; Procedure: Laparoscopic Sleeve Gastrectomy
- Marcaine (Bupivicaine) (Active Comparator): Patient will have Marcaine (Bupivicaine) injected at Laparoscopic Port sites during the Laparoscopic Roux en Y or Laparoscopic Sleeve Gastrectomy.
  Interventions: Procedure: Laparoscopic Roux en Y gastric bypass; Procedure: Laparoscopic Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic Roux en Y gastric bypass — Laparoscopic Roux en Y gastric bypass
Procedure: Laparoscopic Sleeve Gastrectomy — Laparoscopic Sleeve Gastrectomy

SUMMARY:
This study is designed to evaluate the use of bupivacaine liposome 1.3% compared bupivacaine 0.5% in pain control in post-operative laparoscopic bariatric surgery patient The purpose of this study is to evaluate two local anesthetics and determine if there is an advantage of administering one medication compared over the other. The intent is show that one local anesthetic.allows for improved pain control as per the pain scale ratings of the test subjects.

ELIGIBILITY:
Inclusion Criteria:

-Any patient scheduled to undergo Laparoscopic Roux en Y Gastric Bypass or Laparoscopic Gastric Sleeve with Dr. Stephen Fleischer

Exclusion Criteria:

* Patients with an allergy to either medications being studied any patient with neurological disorders that may be exacerbated by the use of either medication,including multiple sclerosis and amyotrophic lateral sclerosis or that may impact the perception of pain.
* Patients with complex medical conditions that may confound data analysis per the principal investigator's discretion.
* Any pregnant patient.Any patients that would not like to participate in the study.
* Any patient that is not able to read or understand English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Subjective Post Operative Pain Level | Within the first 10 days after surgery
  Post operative pain will be assessed on an subjective level. The patient's pain will be assessed by the use of the Wong-Baker pain scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Smith, Principal Investigator — Kettering Health Network

REFERENCES:
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] McGee, DL. Local and topical anesthesia in clinical procedures in Emergency Medicine, 5th edition, Roberts, JR, 263Hedges, JR(Eds), Saunders Elsevier, Philadelphia 2010, pg. 481
- [Background] Weingart SN, Iezzoni LI, Davis RB, Palmer RH, Cahalane M, Hamel MB, Mukamal K, Phillips RS, Davies DT Jr, Banks NJ. Use of administrative data to find substandard care: validation of the complications screening program. Med Care. 2000 Aug;38(8):796-806. doi: 10.1097/00005650-200008000-00004. PMID 10929992
- [Background] Fleischmann KE, Goldman L, Young B, Lee TH. Association between cardiac and noncardiac complications in patients undergoing noncardiac surgery: outcomes and effects on length of stay. Am J Med. 2003 Nov;115(7):515-20. doi: 10.1016/s0002-9343(03)00474-1. PMID 14599629
- [Background] Dimick JB, Chen SL, Taheri PA, Henderson WG, Khuri SF, Campbell DA Jr. Hospital costs associated with surgical complications: a report from the private-sector National Surgical Quality Improvement Program. J Am Coll Surg. 2004 Oct;199(4):531-7. doi: 10.1016/j.jamcollsurg.2004.05.276. PMID 15454134
- See also: CDC — http://cdc.org
- See also: Related Info — http://Uptodate.com